CLINICAL TRIAL: NCT01485523
Title: Sensitivity and Specificity of Nasal Provocation Test in Allergic Rhinitis to House Dust Mites
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 5103
Record Dates: First submitted 2011-12-01; First posted 2011-12-05 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-03

CONDITIONS: Allergic Rhinitis
Keywords: Allergic rhinitis; Nasal provocation test
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Interleukin-13

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients: A = Patients with allergic rhinitis sensitized to dust mites
  Interventions: Other: Nasal provocation test
- Control Subjects: B = control subjects with allergic rhinitis not sensitized to dust mites C = control subjects without allergic rhinitis
  Interventions: Other: Nasal provocation test

INTERVENTIONS:
Other: Nasal provocation test — TPNC to dust mite has an interest in the diagnosis of allergic rhinitis to dust mites when there remains a doubt due to the poly sensitization of the patient, or the lack of specific symptoms and / or the variability of the allergic symptoms during the year. However, this test has not completely validated with a study including a significant number of patients. That's why we plan a prospective single-center comparative open study with the main objective is to determine the sensitivity and specificity of conventional nasal provocation test (TPNC) in 120 patients of 18 to 65 years old with allergic rhinitis sensitized to dust mites and patients with allergic rhinitis not sensitized to dust mites. Our secondary objective is to compare the TPNC a faster TPN-called "minute" (60 minutes) and which allow a wider use. If we demonstrate the validity of TPN then it would become the gold standard needed to decide on a desensitisation to mites.
  Other Names: A patients with allergic rhinitis sensitized to dust mites; B control subjects with allergic rhinitis not sensitized to dust mites; C control subjects without allergic rhinitis

SUMMARY:
The diagnosis of allergic rhinitis to dust mites is difficult and based on three elements : suggestive symptoms of clinical sensitization to dust mites (rhinitis), the existence of an IgE sensitization defined by skin tests and / or specific IgE positive to mite and finally the presence of mite allergens in the environment where the patient is symptomatic. Unfortunately, the link between symptoms and exposure to dust mites is rarely found and according to in the literature, 30% of rhinitis sensitized to house dust mites did not react during a conventional nasal provocation test (TPNC) to dust mites. Thus, TPNC to dust mite has an interest in the diagnosis of allergic rhinitis to dust mites when there remains a doubt due to the poly sensitization of the patient, or the lack of specific symptoms and / or the variability of the allergic symptoms during the year. However, this test has not been completely validated with a study including a significant number of patients. That's why the investigators plan a prospective single-center comparative open study with the main objective is to determine the sensitivity and specificity of conventional nasal provocation test (TPNC) in 120 patients of 18 to 65 years old with allergic rhinitis sensitized to dust mites and patients with allergic rhinitis not sensitized to dust mites. The investigators secondary objective is to compare the TPNC a faster TPN-called "minute" (60 minutes) and which allow a wider use. If the investigators demonstrate the validity of TPN then it would become the gold standard needed to decide on a desensitisation to mites.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking or smoking less than five cigarettes per day
* Subject affiliated with a social security system
* Informed consent signed and dated by the investigator and the subject
* Having been informed about the results of prior medical

Exclusion Criteria:

* Moderate to severe persistent asthma (FEV <70%)
* Treatment:

  * H1 antihistamine (stop for less than 7 days) * Non-steroidal analgesics (stop for less than a week)* Central anti-hypertensive for 4 weeks- Corticosteroids: Nasal (stop for less than 7 days)Oral (if supported by more than 10 mg per day, stopping for less than a week)Intramuscular *Imipramine and other tricyclic treatment (stop for less than a week) *Ketotifen (stop for less than two weeks) *Leukotriene antagonists (stop for less than a week) * Nasal vasoconstrictors (one week)*
* Acute bacterial rhinosinusitis, systemic hypertension, myocardial infarction (<3 months), recent stroke (<3 months), known arterial aneurysm, epilepsy treatment, drug allergy
* Inability to measure a change in flow resistance and intra nasal (nasal obstruction complete)
* History of anaphylaxis to the allergen tested
* Nasal surgery 6-8 weeks before the study
* Subject exclusion period (determined by a previous study or in progress)
* Unable to give informed about the information (subject in an emergency situation, difficulties in understanding the subject)
* Inability to understand the maneuvers of nasal provocation test
* Subject in safeguarding justice, under guardianship
* Pregnancy and lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: From the allergy clinic patients who have a rhinitis and positive skin test to mite or to other aeroallergens or negative skin test
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Jacques Braun, Principal Investigator — Hôpitaux Universitaires de Strasbourg; Frédéric De Blay, Study Director — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Pole de pathologie thoracique.Unité d'allergologie, d'asthmologie et de pathologie respiratoire de l'environnement, Strasbourg, France, France

REFERENCES:
- [Derived] de Blay F, Doyen V, Lutz C, Godet J, Barnig C, Qi S, Braun JJ. A new, faster, and safe nasal provocation test method for diagnosing mite allergic rhinitis. Ann Allergy Asthma Immunol. 2015 Nov;115(5):385-390.e1. doi: 10.1016/j.anai.2015.07.014. Epub 2015 Aug 8. PMID 26265011